CLINICAL TRIAL: NCT06848413
Title: The Impact of an Arabic Educational Video on Reducing Ageism and Promoting Positive Attitudes Toward Older Adults Among Physical Therapists An Application of the PEACE Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Meznah Althubaiti, principal Investigator, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E-24-9163
Record Dates: First submitted 2025-02-16; First posted 2025-02-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Physiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Other: Arabic education video intervention based on the Positive Education about Aging and Contact Experiences (PEACE)

INTERVENTIONS:
Other: Arabic education video intervention based on the Positive Education about Aging and Contact Experiences (PEACE) — This video is designed based on the Positive Education about Aging and Contact Experiences (PEACE), which is suitable for professional medical that is Arabic speaker only.

SUMMARY:
Brief Summary The goal of this experimental study is to determine the effectiveness of implementing an Arabic education video intervention based on the Positive Education about Aging and Contact Experiences (PEACE) model in reducing ageism and anxiety, promoting positive attitudes, and increasing knowledge toward older adults and assessing the effect over time among physical therapists.

The main hypothesis:

The investigators hypothesize that an Arabic educational video intervention based on the PEACE model will significantly reduce ageism and anxiety and increase positive attitudes and knowledge about older adults, and the effectiveness will last over time among physical therapists.

Participants will:

* Complete an initial online survey assessing demographic and professional information, as well as measures of ageism, aging knowledge, anxiety about interactions with older adults, and positive and negative age stereotypes (Time-1).
* Watch a 7-minute Arabic video that includes (1) an animated segment addressing ageism and debunking stereotypes and (2) a live-action segment featuring older adults sharing personal stories to promote intergenerational contact (Time-2).
* Complete an attention check followed by the same outcome measures as in Time-1.
* Complete the same set of outcome measures one week later (Time-3) to assess any changes.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Saudi physical therapists.
* at least one year experience.

Exclusion Criteria:

* Students.
* Intern physical therapists.
* Physical therapy technicians.

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ageism Measure | Baseline in week 1 and after intervention in week 2.
  Ageism was measured using the Fraboni Scale of Ageism (FSA), which was originally developed by Fraboni and revised by Rupp, Vodanovich, and Credé. FSA constitutes a reliable, valid, and multidimensional measure of ageism. Participants will rate 22 items concerning their attitudes toward older adults, from 1 (strongly disagree) to 6 (strongly agree) scale.
Aging Knowledge | Baseline in week 1 and after intervention in week 2.
  Aging knowledge was assessed using the Facts on Aging quiz (FAQ) developed by Palmore's . FAQ is used to measure the basic facts and frequent misconceptions about aging. This measure is valid and has group reliability. In addition, FAQ is currently considered the gold standard. The FAQ is a self-report scale containing 25 questions with a "true" or" false" response and takes less than 5 minutes to complete.
Anxiety about interacting with older adult | Baseline in week 1 and after intervention in week 2.
  Hutchison was developed and tested of the interaction anxiety about older adult measure. This measure assessed participants' feelings of discomfort or anxiety when interacting with older adults. The scale contains 3 items, and the participants will be rating each items concerning their anxiety from 1 (strongly disagree) to 6 (strongly agree).

OTHER OUTCOMES:
Attention Checks | After intervention in week 2.
  Attention checks were designed consistently with to ensure that participants are actively engaged and paying attention after watching the video. Participants will be assigned to respond to 4 attention checks in total. To assess the level of attention after watching the video, the participants will be asked, "Did you watch the video?" (attention checks 1)", and then will be asked, "What was the video you saw about?" (attention check 2), and to assess the participant's comprehension and memory, "please list a thing you remember from the video you were exposed to" (attention checks 3-4). Those who failed to pass a certain threshold (at least two of the four attention checks) will be excluded from the analysis to ensure the reliability of the data collected.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia